CLINICAL TRIAL: NCT02591212
Title: Connecting Through Educational Training: A Pilot of Bystander Training Programming in Sexual Violence and Subtance Abuse
Brief Title: A Pilot of Bystander Training Programming in Sexual Violence and Subtance Abuse
Acronym: P_ConnectED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Heather Bush, Kate Spade & Company Endowed Professor, Associate Professor, Biostatistics, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC R01CE 2690
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Sexual Violence
Keywords: Bystanding behaviors; Campus; Prevention; Sexual Assault; CampusSave

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- #ConnectDots (Active Comparator): Green Dot Intensive Bystander Training (INT Condition) (Randomized):
  Green Dot bystander intervention program (www.livethegreendot.com) seeks to empower potential bystanders (students) to actively engage their peers in violence prevention. Intensive bystander training involves interactive, skill development with role-play of bystander behaviors. This program focuses on building knowledge and skills related to interpersonal violence and being an active bystander. There is a structured curriculum for both introductory sessions and longer, skill-building sessions.
  Administered by: UK VIP Delivery Mode: Class or large groups of 100-150 students; training lasts 3 hours Required: Elective. All students randomized to this condition will be scheduled for training.
  Interventions: Behavioral: Green Dot
- #ConnectWell (Placebo Comparator): Wellness Initiatives for Student Empowerment delivered by UK's Student Wellness Office Programming: Addresses elements of student wellness including campus resources for health issues, AOD abuse prevention/harm reduction strategies, time management and study tips, stress management and reduction, and healthy coping strategies. Training may also provide information on academic resources, money management, and other elements of healthy adaptation to college life.
  Administered by: UK VIP/Student Wellness Ambassadors Delivery Mode: Class or large groups of 100-150 students; training lasts 3 hours Required: Elective. All students randomized to this condition will be scheduled for training
  Interventions: Behavioral: Wellness Initiatives for Student Empowerment

INTERVENTIONS:
Behavioral: Green Dot — Green Dot bystander intervention program (www.livethegreendot.com) seeks to empower potential bystanders (students) to actively engage their peers in violence prevention. Intensive bystander training involves interactive, skill development with role-play of bystander behaviors. This program focuses on building knowledge and skills related to interpersonal violence and being an active bystander. There is a structured curriculum for both introductory sessions and longer, skill-building sessions.
  Arms: #ConnectDots
Behavioral: Wellness Initiatives for Student Empowerment — Wellness training to be provided in modules by Student Wellness ambassadors (http://www.uky.edu/wise). The Student Wellness Ambassadors mission is to inform students on aspects of wellness such as alcohol, drugs, mental health, general well-being, and financial wellness in orer to promote safe and responsible lifestyle decisions. Intervention will address elements of student wellness including campus resources for health issues, AOD abuse prevention/harm reduction strategies, time management and study tips, stress management and reduction, and healthy coping strategies. Training may also provide information on academic resources, money management, and other elements of healthy adaptation to college life.
  Other Names: WISE
  Arms: #ConnectWell

SUMMARY:
The purpose of this randomized intervention pilot is to evaluate the relative efficacy of bystander training elements (delivery mode and integration of substance abuse prevention) among cohorts of incoming undergraduates at the University of Kentucky, a nationally recognized leader in addressing sexual violence through bystander intervention programming. Per university policy, all incoming undergraduates will participate in mandatory online training covering sexual violence awareness, bystander concepts, and alcohol use/abuse. Consenting students will be randomized to one of the following training conditions:

1. Green Dot Intensive Bystander Training (INT) or
2. Student Wellness Training (active control). Students in each condition will be followed for 9 months, one academic year.

DETAILED DESCRIPTION:
Overview: Incoming students will be invited to participate in a randomized pilot testing bystander program efficacy. Those consenting to study participation will be randomized to one of the three conditions. All students are required to take Online sexual violence, bystander and alcohol awareness training (UK mandated HAVEN + Alcohol Edu). Those consenting to study participation will be randomized to one of three conditions: Green Dot (INT) or Student Wellness skills training (active control) provided by UK Student Affairs staff in the Violence Intervention and Prevention Center or the Student Wellness Office. All students agreeing to study participation will be invited to complete surveys at baseline (prior to training), and at 2-3 months after training and 6 months following training (late April, early May). For this pilot, students will be contacted for participation in November of their first year, we anticipate approximately 1,500 students.

Mandatory (UK) Online Training: Alcohol abuse and violence prevention using bystander approach AlcoholEdu: Confidential substance abuse education course which uses a science-based approach to educate students about alcohol and its effects. Whether the student drinks or not, the course will help them make informed decisions about alcohol and better deal with drinking behavior that may occur around them. AlcoholEdu is used by more than 500 colleges nationwide through EVERFi.

Haven provides students with definitions and statistics associated with sexual assault and relationship violence, bystander skills and strategies, and campus policies and resources. The trainings are "personalized and reflective" and incorporate the student's "unique perspectives and experiences." This 45-minute training is mandatory and students are asked to complete a follow-up survey 45-days after the training. Because this training is mandatory for all incoming students, all students are expected to have exposure to this training.

INT Condition (Randomized): Delivered by UK's Violence Intervention and Prevention (see letter from Director Henry):

Green Dot bystander intervention program (www.livethegreendot.com) Programming: Seeks to empower potential bystanders (students) to actively engage their peers in violence prevention. Intensive bystander training involves interactive, skill development with role-play of bystander behaviors. This program focuses on building knowledge and skills related to interpersonal violence and being an active bystander. There is a structured curriculum for both introductory sessions and longer, skill-building sessions. This is currently provided at UK in classrooms, residence halls, etc. Tailored programming is provided to Greek organizations, Living Learning Communities, faculty/staff, etc. While a Popular Opinion Leader strategy13 has been used in prior training, for this trial all incoming students randomized to this condition will be offered intensive bystander training.

Administered by: UK VIP Delivery Mode: Class or large groups of 120-150 students; training lasts 3-4 hours Required: Elective. All students randomized to this condition will be scheduled for training.

NOTE: Green Dot Speeches will be supplemental to Intensive Green Dot Bystander training. Speeches are often given through planned events (UK 101) or students, faculty or staff can request such presentations. These speeches will continue to occur as usual. As the aim of this study is to compare bystander intensive training, we will not attempt to limit participation to Green Dot Speeches.

Training Control Condition (Randomized): Delivered by UK's Student Wellness Office (Drew M. Smith) Programming: Addresses elements of student wellness including campus resources for health issues, AOD abuse prevention/harm reduction strategies, time management and study tips, stress management and reduction, and healthy coping strategies. Training may also provide information on academic resources, money management, and other elements of healthy adaptation to college life.

Administered by: UK VIP Delivery Mode: Class or large groups of 120-150 students; training lasts 3-4 hours Required: Elective. All students randomized to this condition will be scheduled for training.

General Statistical Considerations. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation, median, first and third quartiles, and min and max); categorical variables will be described with counts and percentages. Change scores and percent change scores will be calculated from baseline for follow-ups at 4- and 9-months. Numerical and graphical summaries will be provided overall, by subpopulation within college communities (e.g., by gender, sexual attraction, fraternity/sorority or athletic team membership) and most importantly by training condition. Simple comparisons of groups will be made using ANOVA for continuous variables and chi-square tests for categorical outcomes. Comparisons between groups will be conducted as randomized; simple comparisons of continuous variables between groups will be performed using ANOVA and chi-square tests of independence for categorical variables. Although groups will be randomly assigned, potential confounders will be examined with bivariate analyses and comparisons requiring covariate adjustment will use regression modeling (e.g. ANCOVA, logistic regression).

Analysis Plan: The primary purpose of the pilot is to determine feasibility and to examine strategies for recruiting and training students. However, the primary analysis is the as randomized comparison of the cumulative reports of bystanding behaviors collected during the academic year between the two training conditions. A one-way ANOVA (with corresponding post-hoc tests to compare specific groups) will be used to compare the primary outcome of bystander behaviors (measured as the sum of frequency responses to bystander behaviors over the academic year) between those randomzied to INT versus SubINT conditions. Analyses will be conducted without adjustment, adjusting only for academic year, and adjusting for potential confounders not controlled for by randomization. Secondary outcomes will also be compared using a one-way ANOVA. A two-sided significance level of 0.01 will be used to protect against a Type I error in the presence of multiple comparisons. Post-hoc comparisons of groups will only be conducted when the overall F-test suggests differences between groups. All analyses for primary outcomes for will be conducted using comparison groups as randomized for an intent-to-treat (ITT) analysis. For those who are lost to follow-up, multiple imputation will be used in the ITT analysis. Sensitivity analyses using as observed data and single imputation (LOCF) will also be conducted. We will also perform analyses using a modified ITT (mITT), where participants electing not to pursue the intensive training are excluded, but groups are still compared as randomized. The primary analysis is the longitudinal analyses will be conducted using linear mixed models (PROC MIXED) to investigate differences between conditions, trends over time, and whether the time trends differ between conditions. Longitudinal analyses will be conducted by academic year but academic years will also be combined. For combined academic years, the time variable will be included with respect to the online training and academic year will be investigated as a potential confounder. Planned subgroup analyses include analyses by gender group, by sexual attraction, by Greek life participation. These will also be conducted as randomized and as received. Effect modification will also be assessed by including interactions in regression models (linear, logistic, and mixed models depending on outcomes and the presence of longitudinal measures). Participation and completing non-mandatory trainings will be examined overall and by subgroup as well. SAS v9.4 will be used for all data management and statistical analysis; a significance level of 0.01 will be used for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

-Incoming University of Kentucky undergraduate students (2015)

Exclusion Criteria:

* Any current/non-incoming University of Kentucky student
* Any student primarily enrolled at another college or university

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 427 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Bystanding Behaviors increase bystander efficacy and behaviors by domain (alcohol abuse and violence prevention). | One academic year (9 months)
  The primary outcome for this study is bystanding behaviors as measured by the number of behaviors reported by students overall and by domain. Bystanding behaviors are measured through reports of actual behaviors. These primary bystanding behavior outcomes will be used to evaluate the relative efficacy of the intervention(s). As bystanding requires opportunity, these primary outcomes will be examined accounting for the presence of opportunity to bystand. The primary analysis will be the comparison of these outcomes over time using mixed models, with a particular interest on whether there is a condition by time interaction (time: baseline, 3 months post, 6 months post).
Bystanding Behavior Intentions Scale | One academic year (9 months)
Bystanding Behavior Efficacy Scale | Academic Year (9 months)
Bystanding Behaviors Engagement with Peers Scale | Academic Year (9 months)

SECONDARY OUTCOMES:
Acceptance of SV/DV Scale | One academic year (9 months)
Number of risky behaviors, sexual and alcohol related | One academic year (9 months)

OTHER OUTCOMES:
Social media and campus communications (e.g., Twitter, Instagram, Facebook, myUK app, text messaging features). | One academic year (9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Bush, PhD, Principal Investigator — University of Kentucky; Ann L Coker, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States